CLINICAL TRIAL: NCT01428921
Title: Long-term Efficacy of Extended Education Programme on Improving Treatment Adherence to Continuous Positive Airway Pressure in Obstructive Sleep Apnea
Brief Title: Long Term Efficacy of Education Programme on Continuous Positive Airway Pressure Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lai Yuen Kwan Agnes, Senior Technical Officer, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UW11-044
Record Dates: First submitted 2011-09-01; First posted 2011-09-05 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-10

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Long-term efficacy; Education programme; Adherence; OSA; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extended Education (Experimental): * Standard education programme as described above,
  * Plus
    1. Face-to-face session (Part 1: Knowledge Enhancement Session, Part 2: Brief Motivation Interview Session) after the morning of CPAP titration
    2. Follow-up phone call would be arranged within 1 week after using CPAP.
    3. Video, slides and booklets would be used as education media.
  Interventions: Behavioral: Theory based education and brief motivation interview
- Standard education (No Intervention): - Each subject will receive advice from Sleep Lab staff on the need for CPAP treatment, and the care of CPAP device and mask.

INTERVENTIONS:
Behavioral: Theory based education and brief motivation interview — * Standard education programme as described above,
  * Plus
    1. Face-to-face session (Part 1: Knowledge Enhancement Session, Part 2: Brief Motivation Interview Session) after the morning of CPAP titration
    2. Follow-up phone call would be arranged within 1 week after using CPAP.
    3. Video, slides and booklets would be used as education media.
  Other Names: Education program; CPAP adherence
  Arms: Extended Education

SUMMARY:
Obstructive sleep apnea (OSA) is a common sleep disorders associated with excessive daytime sleepiness and cardiovascular disease. Continuous positive airway pressure (CPAP) therapy is an effective standard treatment and is widely prescribed for patients with OSA. Successful CPAP treatment has also been shown to improve cognitive, cardiovascular and metabolic function. Sustainable CPAP treatment would alleviate the substantial cost burden of health-related consequences of untreated OSA.

However, the use of CPAP for such patients is disappointingly low and limits the effectiveness of treatment. Early CPAP education and follow up have shown to be very important in helping subjects to handle side-effects or problems associated with the use of CPAP. Good education program at the initial phase of using CPAP is essentially affected the acceptance and adherence of CPAP therapy. Good CPAP adherence is not only medically essential to patients' health but also economically importance to society by alleviating the substantial cost burden of health-related consequences.

To the best of our knowledge, there is no randomized clinical trial (RCT) to prove the long-term efficacy of extended education program on improving continuous positive airway pressure use and its treatment outcomes.

The primary purpose of this study is to assess the long-term efficacy of our on-going RCT which is an extended education program on improving CPAP compliance.

The investigators hypothesize that the application of both MI technique and SCT-based extended education program at the initial phase of using CPAP also would enhance CPAP adherence even after one year of attending education class.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common disease characterized by recurrent episodic collapse of the upper airway during sleep. It affects 4-5% of the middle-aged population. Continuous positive airway pressure (CPAP) is an effective treatment to relieve the repetitive upper airway obstruction during sleep, and to improve cognitive, cardiovascular and metabolic function. However, compliance to CPAP treatment has been less than ideal which limits its effectiveness.

Sustained CPAP treatment would alleviate the substantial cost burden of health-related consequences of untreated OSA. Early CPAP education and follow up have been shown to be very important in helping subjects to handle side-effects or problems associated with the use of CPAP. However, all current randomized controlled trials only evaluated its short-term efficacy for not more than 6months. Only one retrospective observational study assessed the longer term (1 year) effect of an education program by assessing patients' re-attendance rate of CPAP clinic. However, this study suffers from the residual effects of confounders. Therefore, the investigators need long term assessment of education program on CPAP compliance based on properly conducted randomized control trial.

Our team has developed a theory-based behavioral education program to improve CPAP compliance. It utilizes social cognitive theory (SCT) and motivation interviewing (MI) which are popularly used theory-based education strategies and have been widely adopted and shown to be more effective than the traditional approach in health education programs. However, such programs have not been examined the longer term effect of education program in OSA patients. The investigators have recently started a RCT that assesses the 3-month effect of the program. To date, the investigators have recruited 36 subjects in 5 months. The subject recruitment is conservatively expected to be completed by July 2011. By the time when the review process of this proposal is completed, most of these subject should have been on treatment by 1 year. Hence, it is very timely for us to catch up this group of subjects for assessing the long-term effect of our education program.

In additional, our team is highly experienced in the management of OSA patients. The investigators have recently demonstrated that the use of CPAP on the improvement cardiovascular and metabolic functions. Currently, the investigators are conducting a randomized controlled trial "Education and CPAP" (IRB no. UW10-177)(NCT01173406), which is to assess the short-term (3-months) efficacy of extended education program, which uses the concepts of SCT and MI.

To the best of our knowledge, there is no randomized study from other investigators on the long-term efficacy of CPAP education intervention (either using traditional or theory-based education strategy). This proposed study is to assess the long-term efficacy of our current on-going extended education program on improving CPAP compliance on Chinese subjects with OSA.

ELIGIBILITY:
Inclusion Criteria:

-All 100 subjects recruited in our on-going RCT (IRB no. UW10-177)(ClinicalTrials.gov identifier no. NCT01173406) will be invited to participate in this extended study.

Exclusion Criteria:

-Unable to obtain the written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
CPAP usage | 1 year after recieving CPAP education
  It is to assess objective CPAP usage at 1 year after receiving CPAP education.

SECONDARY OUTCOMES:
To evaluate the treatment outcomes of CPAP therapy on neuropsychologic aspects | at 1 year after recieving CPAP education
  To evaluate the treatment outcomes of CPAP therapy on neuropsychologic aspects such as the change in Epworth Sleepiness Score

CONTACTS AND LOCATIONS:
Overall Officials: Agnes YK Lai, MSc, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong, Hong Kong